CLINICAL TRIAL: NCT06202248
Title: A Feasibility and Safety Study of Focal Interstitial Radiotherapy Using Diffusing Alpha Emitters Radiation Therapy (DaRT) Seeds in Men With Non-metastatic Locally Recurrent Prostate Cancer.
Brief Title: A Study to Assess Alpha DaRT224 for the Treatment of Men With Non-metastatic Locally Recurrent Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-PRST-00
Record Dates: First submitted 2023-12-31; First posted 2024-01-11 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-05

CONDITIONS: Non-metastatic Prostate Cancer; Locally Recurrent Prostate Cancer
Keywords: recurrent prostate cancer.; Alpha emitting radiation; Alpha DaRT; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DaRT Seeds (Experimental): Intratumoral Diffusing alpha-emitters Radiation Therapy (DaRT) Seeds
  Interventions: Device: Experimental: DaRT seeds

INTERVENTIONS:
Device: Experimental: DaRT seeds — Intratumoral Diffusing alpha-emitters Radiation Therapy (DaRT) Seeds

SUMMARY:
This is a multi-center clinical study enrolling up to 10 participants. The purpose of this study is to assess the feasibility and safety of intratumoral DaRT seeds implantation for the treatment of locally recurrent prostate cancer. Secondary objectives are to 1. To evaluate feasibility of interstitial radiotherapy using DaRT seeds.

Feasibility will be determined according to the rate of successful placement of DaRT seeds via imaging [Timeframe: immediately following the insertion procedure 2. To assess the impact of DaRT seeds on patient reported quality of life.

DETAILED DESCRIPTION:
This study is a prospective multicenter, single arm, open label , interventional clinical study to assess the feasibility and safety of intratumoral Alpha DaRT seeds for the treatment of men with non metastatic locally recurrent prostate cancer.

Diffusing Alpha emitters Radiation Therapy (DaRT). Treatment will be delivered through radioactive sources [Ra-224 containing Stainless steel 316LVM tubes- (Alpha DaRT seeds)] inserted into the tumors.

The purpose of this study is to assess the feasibility and safety of intratumoral DaRT seeds implantation for the treatment of locally recurrent prostate cancer. The secondary objectives is 1. To evaluate feasibility of interstitial radiotherapy using DaRT seeds.

Feasibility will be determined according to the rate of successful placement of DaRT seeds via imaging [Timeframe: immediately following the insertion procedure 2. To assess the impact of DaRT seeds on patient reported quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally recurrent prostate adenocarcinoma cancer confined to at least 1 hemi-gland with concordant pathology and imaging findings within 6 months prior to consenting
* Targetable lesion by either PSMA PET-CT according to PERCIST v1.0 or by multiparametric MRI according RECIST v1.1
* Patient being considered for focal salvage brachytherapy
* Lesion size ≤ 3 cm in the longest diameter
* Target lesion technically amenable for full tumor coverage with the Alpha DaRT seeds
* Pre-salvage PSA level (rPSA) below <10 ng/ml
* Age ≥ 18 years old
* ECOG Performance Status Scale ≤ 2
* Subjects' life expectancy is more than 6 months
* Negative metastatic workup on at least standard imaging (CT CAP and bone scan). Other metastatic screening studies allowed in lieu of standard imaging including multiparametric MRI prostate/whole body, PSMA PET, F18 PET or Axumin PET within 3 months before visit 0
* Platelet count ≥100,000/mm3
* Subjects are willing and able to sign an informed consent form.

Exclusion Criteria:

* N1 or M1 disease
* Prior TURP or prostate surgery
* Inability to undergo multiparametric MRI (i.e. permanent implanted device incompatible with MRI)
* Inability to undergo general or spinal anesthesia
* Prior androgen deprivation therapy or systemic chemotherapy for prostate cancer within 3 months before visit 0.
* Previous diagnosis of other malignancy < 3 years of enrollment (excluding non-melanomatous skin cancer)
* Volunteers participating in another interventional study in the past 30 days which might conflict with the endpoints of this study or the evaluation of response or toxicity of DaRT
* High probability of protocol non-compliance (in opinion of investigator)
* Subjects not willing to sign an informed consent
* Patients with significant comorbidities that the treating physician deems may conflict with the endpoints of the study (e.g., poorly controlled autoimmune diseases, vasculitis, etc.)

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of intratumoral DaRT seeds implantation | immediately following the insertion procedure
  To evaluate feasibility of interstitial radiotherapy using DaRT seeds. Feasibility will be determined according to the rate of successful placement of DaRT seeds via imaging

CONTACTS AND LOCATIONS:
Overall Officials: Tomer Charas, MD, Principal Investigator — Radiotherapy unit at Rambam Health Care Campus, Israel
Locations (1):
- RAMBAM Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No